CLINICAL TRIAL: NCT06486142
Title: EGFR-mutated Lung Cancer in Randomized Investigator-Initiated Study
Acronym: ERIS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Swedish Lung Cancer Study Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-003755-41
Record Dates: First submitted 2024-05-07; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; EGFR; Osimertinib; Afatinib; Dacomitinib; ctDNA; Resistance mechanisms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; dacomitinib; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Afatinib/Dacomitinib (Active Comparator)
  Interventions: Drug: Afatinib/Dacomitinib
- Osimertinib (Active Comparator)
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Afatinib/Dacomitinib — Second-generation EGFR-inhibitors
  Other Names: Study participants receiving afatinib or dacomitinib until tumor progression/other reasons
  Arms: Afatinib/Dacomitinib
Drug: Osimertinib — Third-generation EGFR-inhibitor
  Other Names: Study participants receiving osimertinib until tumor progression/other reasons
  Arms: Osimertinib

SUMMARY:
The purpose of this study is to evaluate the optimal sequence of EGFR-inhibitors in lung cancer patients with EGFR-positive tumors not amenable for curative treatment. Life quality, adverse effects and tumor response will be evaluated and analyses of obtained blood and tumor samples will be performed to identify molecular profiles and biomarkers that can be used for treatment decisions.

DETAILED DESCRIPTION:
ERIS is an investigator-initiated randomized phase III trial. Non-small cell lung cancer (NSCLC) patients with advanced disease, not amenable for curative treatment, are considered for targeted therapy. For first-line treatment in patients with EGFR-positive tumors there are now several options, of which osimertinib (a third generation EGFR-TKI) and dacomitinib/afatinib (second generation EGFR-TKIs) are considered first-hand choices. Dacomitinib/afatinib treatment might be switched to osimertinib in the event of treatment failure, provided that an EGFR T790M mutation is detected. However, in about half of patients with second generation EGFR- TKI treatment failure, the resistance mechanism is different from T790M. Thus, there is a need to identify which patients that benefit from osimertinib in first line and which patients that rather benefit from a second-generation EGFR-TKI in first line, respectively. Early treatment prediction and monitoring through biomarkers in blood and tumor could be one step forward in individualized treatment.

After being informed about the study patients with EGFR-positive NSCLC, considered for first-line treatment, will sign a consent and undergo a screening period to determine eligibility for study entry. When screening is completed, and inclusion criteria are met, study participants will be randomized in a 1:1 ratio to osimertinib or afatinib/dacomitinib.

Patients randomized to afatinib/dacomitinib will be able to cross-over to osimertinib in the event of progression and confirmed T790M-mutation. In the event of progression on osimertinib or on afatinib/dacomitinib without T790M, the study participants will be treated as chosen by the investigator and in accordance with applicable national guidelines.

Longitudinal blood samples and, when appropriate, tumor tissue/cytology or other fluids (pleural effusion etc.) will be assembled and used for comprehensive analysis to study potential biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* The subject has given written consent to participate in the study.
* Histological or cytological diagnosis of NSCLC.
* Clinical stage III/IV disease (with or without CNS metastasis) or a recurrence not amenable for curative treatment intention.
* Measurable disease according to RECIST 1.1 criteria or equivalent/modified criteria.
* Any WHO PS.
* Age ≥ 18 years, no upper age limit.
* EGFR-mutation in tumor (in cases where tumor tissue is not available for mutation analysis, circulating tumor-DNA (ctDNA) in plasma may serve as inclusion criteria), which is presumably predictive of sensitivity to EGFR TKI.
* Treatment-naive with regard to TKI's
* Negative pregnancy test (blood or urine test)
* For fertile participants, adequate contraception should be used; intrauterine device, bilateral tubal occlusion, vasectomy or abstinence (a reduced effect of hormonal contraception methods due to the drugs cannot be excluded). Pregnancy should be avoided during treatment and the first 4 months following treatment discontinuation.

Exclusion Criteria:

* Condition incompatible with the study or with the planned treatment.
* Present (not radically treated/no planned radical treatment of) other primary malignancy with metastatic potential.
* Co-enrolment in other interventional trial if incompatible with ERIS according to investigator (e.g. due to potential drug interactions).
* Intake of hypericum perforatum (intake must be interrupted before start of study treatment).
* All subjects should avoid concomitant use of medications with known interaction with planned treatment, whenever feasible. If the administration of a medication interacts with any of the three investigational treatments and cannot be exchanged or managed in order to avoid interactions the patient is excluded from the trial.

  * Drugs that can either increase or decrease the concentration of osimertinib in plasma:

    * Strong activators of CYP3A. Simultaneous administration should be avoided.
    * Regular CYP3A4-inhibitors should be used with caution or be avoided.
  * Drugs that can either increase or decrease the concentration of afatinib in plasma:

    * Strong inhibitors of P-glycoprotein should not be administered simultaneously with afatinib, instead it should preferably be 6-12 hours between.
    * Strong activators of P-glycoprotein may reduce exposure of afatinib
  * Drugs that can either increase or decrease the concentration of dacomitinib in plasma:

    * Proton pump inhibitors should be avoided.
    * Simultaneous administration of drugs that are metabolized by CYP2D6 should be avoided. If simultaneous use of that kind of medications are considered necessary, dose recommendations for simultaneous use of respective drug should be followed.
* Any evidence of severe or uncontrolled systemic diseases which in the investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol. Screening for chronic conditions is not required.
* Gastrointestinal conditions incompatible with swallowing or precluding absorption of the study drug.
* Pregnancy or refusal to use contraceptives.
* Abnormal findings of blood chemistry not compatible with the study drug according to investigator.
* History of hypersensitivity to the study drug (or drugs with a similar chemical structure or class) or any excipients.
* Severe hepatic impairment/renal function incompatible with study drug according to investigator.
* Hereditary conditions with galactose intolerance, total lactase deficiency or glucose -galactose malabsorption.
* Congenital long QT syndrome.
* Judgment by the investigator that the subject should not participate in the study, e.g., if the subject is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Maximum 6 years

SECONDARY OUTCOMES:
Time on TKI-treatment | Maximum 6 years
Objective response rate | Maximum 6 years
Disease control rate | Maximum 6 years
Overall survival | Maximum 6 years
Quality of life | Maximum 6 years
  Points on the Lung Cancer Symptom Scale (LCSS) will be compared between the two treatment arms
Hereditary genetic alterations | Within 15 years from end of study
  The frequency of germline DNA variants will be studiedassociated with cancer predisposition will be investigated
Identification of potential blood-borne biomarkers of treatment prediction and resistance | Within 15 years from end of study

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne university hospital, Lund, Sweden